CLINICAL TRIAL: NCT03624036
Title: A Phase 1 Multicenter Study Evaluating the Safety and Tolerability of KTE-X19 in Adult Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: Study to Evaluate the Safety and Tolerability of Brexucabtagene Autoleucel (KTE-X19) in People With Relapsed/Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Acronym: ZUMA-8
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-108; 2018-001923-38 (EudraCT Number)
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia and Relapsed/Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — brexucabtagene autoleucel; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with relapsed/refractory (r/r) chronic lymphocytic leukemia (CLL) will receive conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-cluster of differentiate 19 (CD19) chimeric antigen receptor (CAR) T cells/kg on Day 0.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r CLL will receive conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r CLL and small lymphocytic lymphoma (SLL) with ≤1% malignant cells in peripheral blood or absolute lymphocyte count (ALC) < 5,000 cells/μL will receive conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg on Day 0.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r CLL who previously received two lines of therapy along with ibrutinib with or without anti CD20 antibodies, B-cell lymphoma 2 (BCL-2) and Phosphoinositide 3-kinase (PI3k) inhibitors will receive ibrutinib up to 30 hours prior to leukapheresis along with conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg on Day 0.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Second Stage Cohort 4B: 2 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r CLL who previously received two lines of therapy along with ibrutinib with or without anti CD20 antibodies, BCL-2 and PI3k inhibitors will receive ibrutinib up to 30 hours prior to leukapheresis along with conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0.
  Upon completion of Cohort 4A, it was determined not to enroll participants in Cohort 4B.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: brexucabtagene autoleucel — CAR-transduced autologous T cells administered intravenously
  Other Names: KTE-X19
Drug: Fludarabine — Administered intravenously
Drug: Cyclophosphamide — Administered intravenously

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of brexucabtagene autoleucel (KTE-X19) in adults with relapsed/refractory chronic lymphocytic leukemia (r/r CLL) and small lymphocytic lymphoma (r/r SLL) who have received at least 2 prior lines of treatment, one of which must include a Bruton's tyrosine kinase (BTK) inhibitor.

After the end of KTE-C19-108, participants who received an infusion of brexucabtagene autoleucel will complete the remainder of the 15-year follow-up assessments in a separate Long-term Follow-up study, KT-US-982-5968 (NCT05041309).

ELIGIBILITY:
Key Inclusion Criteria:

* Documentation of relapsed or refractory CLL and SLL; must have received at least 2 prior lines of treatment, one of which must include a Bruton's tyrosine kinase (BTK) inhibitor.

  * Cohort 1 and 2: Participants with r/r CLL who have received at least 2 prior lines of treatment, one of which must include a BTK inhibitor.
  * Cohort 3: Participants with r/r CLL and SLL must present with ≤ 1% circulating tumor cells in peripheral blood or absolute lymphocyte count (ALC) < 5000 cells/μL. Participants must have received at least 2 prior lines of treatment, one of which must include a BTK inhibitor.
  * Cohort 4: Participants with r/r CLL who have received at least 2 prior lines of treatment and must have received ibrutinib as a single agent or in comibation with anti-cluster of differentiate 20 (CD20) antibodies, B-cell lymphoma 2 (BCL-2) inhibitors, and phosphoinositide 3-kinase inhibitor (PI3k) inhibitors for at least 6 months as the last line of therapy prior to screening. Ibrutinib administration will continue up to 30 hours prior to leukapheresis. In case of treatment interruption with ibrutinib, the principal investigator should reach out to the medical monitor to discuss.
* An indication for treatment per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria and radiographically measurable disease (at least 1 lesion > 1.5 cm in diameter)
* Adequate hematologic function as indicated by:

  * Platelet count ≥ 50 × 10^9/L
  * Neutrophil count ≥ 0.5 × 10^9/L
  * Hemoglobin ≥ 8 g/dL unless lower values are attributable to CLL
* Adequate renal, hepatic, cardiac and pulmonary function defined as:

  * Creatinine clearance (as estimated by Cockcroft-Gault) ≥ 60 mL/min
  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 mg/dL unless participant has Gilbert's syndrome
  * Left ventricular ejection fraction (LVEF) ≥ 50%, no evidence of pericardial effusion, no New York Heart Association (NYHA) class III or IV functional classification, no clinically significant arrhythmias
  * No clinically significant pleural effusion
  * Baseline oxygen saturation > 92% on room air
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy or BTKi (ibrutinib or acalabrutinib) at the time the participant is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy. At least 3 half-lives must have elapsed from any prior systemic inhibitory/stimulatory immune checkpoint molecule therapy at the time the participant is planned for leukapheresis (eg, ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists)

Key Exclusion Criteria:

* A history of treatment including any of the following:

  * Prior cluster of differentiate 19 (CD19) directed therapy
  * Prior allogeneic hematopoietic stem cell transplant (SCT) or donor lymphocyte infusion (DLI) within 6 months prior to enrollment
* History of autoimmune disease resulting in end-organ injury unless attributable to CLL (eg, idiopathic thrombocytopenic purpura (ITP), autoimmune hemolytic anemia (AIHA))
* Diagnosis of Richter's transformation or a history of malignancy other than non-melanoma skin cancer or carcinoma in situ (eg, skin, cervix, bladder, breast), superficial bladder cancer, asymptomatic localized low grade prostate cancer for which watch-and-wait approach is standard of care, or any other cancer that has been in remission for > 3 years prior to enrollment
* History of severe hypersensitivity reaction attributed to aminoglycosides

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (22):
- United States (21):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Stanford, California
  - Sarah Cannon - Denver, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Center, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Cancer Hospital, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davids MS, Kenderian SS, Flinn IW, Hill BT, Maris M, Ghia P, et al. ZUMA-8: A Phase 1 Study of KTE-X19, an Anti-CD19 Chimeric Antigen Receptor (CAR) T-Cell Therapy, in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia. Blood. 2022;140:7454-6.
- [Derived] Davids MS, Kenderian SS, Flinn I, Hill BT, Maris M, Ghia P, Byrne M, Bartlett NL, Pagel JM, Zheng Y, Kanska J, Zhang W, Granados E, Pinilla-Ibarz J. ZUMA-8: a phase 1 study of brexucabtagene autoleucel in patients with relapsed/refractory chronic lymphocytic leukemia. Blood. 2025 Aug 21;146(8):938-943. doi: 10.1182/blood.2024027460. PMID 40209059
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Italy. The study was terminated before enrolling participants in the Cohort 4B.
Pre-assignment Details: 17 participants were screened.
Groups:
- First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with relapsed/refractory (r/r) chronic lymphocytic leukemia (CLL) received conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered intravenously (IV) on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-cluster of differentiate 19 (CD19) chimeric antigen receptor (CAR) T cells/kg administered IV on Day 0.
- First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r CLL received conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered IV on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 2 x 10^6 anti-CD19 CAR T cells/kg administered IV on Day 0.
- Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r CLL and small lymphocytic lymphoma (SLL) with ≤1% malignant cells in peripheral blood or absolute lymphocyte count (ALC) < 5,000 cells/μL received conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered IV on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg administered IV on Day 0.
- Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r CLL who previously received two lines of therapy along with ibrutinib with or without anti CD20 antibodies, B-cell lymphoma 2 (BCL-2) and Phosphoinositide 3-kinase (PI3k) inhibitors received ibrutinib up to 30 hours prior to leukapheresis along with conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered IV on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg administered IV on Day 0.
Period: Overall Study
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Started | 7 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 3 | 3 | 3
Not completed — Death | 2 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Enrolled but Never Treated | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 3 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were treated with any dose of brexucabtagene autoleucel.
Groups:
- First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r CLL received conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered IV on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg administered IV on Day 0.
- Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r CLL and SLL with ≤1% malignant cells in peripheral blood or ALC < 5,000 cells/μL received conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered IV on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg administered IV on Day 0.
- Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r CLL who previously received two lines of therapy along with ibrutinib with or without anti CD20 antibodies, BCL-2 and PI3k inhibitors received ibrutinib up to 30 hours prior to leukapheresis along with conditioning chemotherapy (fludarabine 30 mg/m^2/day over 30 minutes and cyclophosphamide 500 mg/m^2/day over 30-60 minutes) administered IV on Days -5 to -3 with 2 rest days, followed by single infusion of brexucabtagene autoleucel 1 x 10^6 anti-CD19 CAR T cells/kg administered IV on Day 0.
- Total: Total of all reporting groups
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 1 | 1 | 9
  >=65 years | 2 | 0 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (5.8) | 58.7 (5.9) | 68.0 (11.5) | 63.3 (9.1) | 62.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 1 | 5
  Male | 3 | 2 | 3 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 3 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 5 | 3 | 3 | 2 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 2 | 3 | 3 | 14
  Italy | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: DLTs refer to toxicities with onset experienced during the first 28 days of study treatment that have been judged to be clinically significant and related to study treatment. DLTs evaluated may include with some exceptions: All brexucabtagene autoleucel related Grade 3 non-hematologic toxicities lasting for more than 7 days, Grade 4 non-hematologic toxicities regardless of duration, and Grade 4 hematologic toxicity lasting more than 30 days if not attributable to underlying disease.
Time Frame: First infusion date of brexucabtagene autoleucel up to 28 days. Participants were evaluated in specified period but Grade 4 hematologic toxicity (specified in description) having onset in this period were further observed for 30 days for confirmation.
Population: DLT Evaluable Set included all participants treated with the target brexucabtagene autoleucel dose and followed for at least 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 6 | 3 | 3 | 3
Participants | 0 | 0 | 1 | 0

2. Secondary Outcome: Objective Response Rate (ORR) Per Investigator Review Assessed by International Workshop on CLL (IWCLL) 2018 Criteria
Description: ORR was defined as percentage of participants achieving either complete response (CR), complete response with incomplete hematopoetic recovery (CRi) or partial response (PR). Criteria for CR: no lymphadenopathy >1.5 cm or hepatomegaly/splenomegaly, lymphocytes <4000/microliters (μL), bone marrow sample must be normocellular with 30% lymphocytes and no B-lymphoid nodules, platelets ≥100,000/µL, hemoglobin ≥11 grams per deciliter (g/dL). CRi: All CR criteria were met except with platelet count <100,000/μL, hemoglobin <11 g/dL or neutrophil count <500/μL. PR: ≥1 of these: ≥50% decrease in lymphocytes, lymphadenopathy, size of liver and spleen, 50% decrease in bone marrow infiltrates; and ≥1 of these: platelets ≥100,000/µL or ≥50% increase from Baseline, hemoglobin ≥11 g/dL or ≥50% increase from Baseline. Participants who did not meet criteria were considered nonresponders. 95% confidence interval (CI) was calculated by Clopper-Pearson method.
Time Frame: First infusion date up to last follow up visit (maximum duration: 42 months)
Population: All Treated Subjects Set included all participants who were treated with any dose of brexucabtagene autoleucel.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 6 | 3 | 3 | 3
percentage of participants | 50 [11.8 to 88.2] | 33 [0.8 to 90.6] | 100 [29.2 to 100.0] | 0 [0.0 to 70.8]

3. Secondary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant that does not necessarily have a relationship with study treatment or worsening of a pre-existing medical condition. TEAEs were defined as AEs with onset on or after the initiation of brexucabtagene autoleucel infusion.
Time Frame: First infusion date up to last follow up visit (maximum duration: 42 months)
Population: Safety Analysis Set included all participants who were treated with any dose of brexucabtagene autoleucel.
Measure: Number; unit: percentage of participants
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 6 | 3 | 3 | 3
percentage of participants | 100 | 100 | 100 | 100

4. Secondary Outcome: Peak Level of Anti-CD19 CAR T-Cells in Blood
Description: Peak was defined as the maximum number of CAR T cells measured post-infusion.
Time Frame: First infusion date up to 3 months post-infusion (approximately 3 months)
Population: Participants in the safety analysis set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: cells/μL
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 6 | 2 | 3 | 3
cells/μL | 1.46 [0.58 to 2.35] | 1.08 [0.00 to 2.15] | 42.18 [27.52 to 679.38] | 1.00 [0.00 to 1.27]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to last follow up visit (maximum: 43 months); Adverse Events: First infusion date up to last follow up visit (maximum: 42 months)
Description: All-Cause Mortality: All Enrolled Analysis Set included all the enrolled participants.
  Adverse Events: Safety Analysis Set included all participants who were treated with any dose of brexucabtagene autoleucel.
Arm/Group | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg
All-Cause Mortality (participants affected / at risk) | 2/7 | 3/3 | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/3 | 3/3 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=6) | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg (N=3) | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=3) | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=3)
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | First Stage Cohort 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=6) | First Stage Cohort 2: 2 x 10^6 Anti-CD19 CAR T Cells/kg (N=3) | Second Stage Cohort 3: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=3) | Second Stage Cohort 4A: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 3 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 1 | 1 | 2
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 2 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0
Frustration tolerance decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03624036/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT03624036/SAP_001.pdf
  • Statistical Analysis Plan: Translational Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT03624036/SAP_002.pdf